CLINICAL TRIAL: NCT01401374
Title: Online Health Survey of Patients With Vitiligo Vulgaris/ Online Survey of Pediatric Patients With Vitiligo
Status: Completed | Type: Observational
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Sponsor
Other Study IDs: 10-148/10-149x
Record Dates: First submitted 2011-07-21; First posted 2011-07-25 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Vitiligo Vulgaris
Keywords: Vitiligo Vulgaris; Autoimmunity; Thyroid Disease
MeSH Terms: conditions — Vitiligo; Autoimmune Diseases; Thyroid Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Vitiligo Patients: patients with vitiligo vulgaris
- Controls: Individuals without vitiligo vulgaris

SUMMARY:
The study is an on-line survey posted on survey monkey that addresses some demographic and environmental issues that could potentially relate to vitiligo vulgaris onset or disease exacerbation.

DETAILED DESCRIPTION:
The survey is designed to look at some issues that are pertinent to individuals with vitiligo, including access to care, severity of disease, under-reported disease activity, causative and exacerbating factors and co-morbid illnesses.

ELIGIBILITY:
Inclusion Criteria:

* Ability to complete survey

Exclusion Criteria:

* Inability to complete survey

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals self-reporting vitiligo vulgaris and controls who do not have vitiligo vulgaris
Sampling Method: Non-Probability Sample
Enrollment: 3258 (Actual)
Dates: Start 2011-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Correlation of Disease State in Vitiligo with Clinical and Psychological Measures | Self-reported retrospective single survey

CONTACTS AND LOCATIONS:
Overall Officials: Nanette Silverberg, MD, Principal Investigator — St. Luke's-Roosevelt Hospital Center
Locations (1):
- St. Luke's-Roosevelt Hospital Center, New York, New York, United States

REFERENCES:
- [Derived] Silverberg JI, Reja M, Silverberg NB. Regional variation of and association of US birthplace with vitiligo extent. JAMA Dermatol. 2014 Dec;150(12):1298-305. doi: 10.1001/jamadermatol.2014.899. PMID 25006795
- [Derived] Silverberg JI, Silverberg NB. Quality of life impairment in children and adolescents with vitiligo. Pediatr Dermatol. 2014 May-Jun;31(3):309-18. doi: 10.1111/pde.12226. Epub 2013 Oct 18. PMID 24304125
- [Derived] Silverberg JI, Silverberg NB. Association between vitiligo extent and distribution and quality-of-life impairment. JAMA Dermatol. 2013 Feb;149(2):159-64. doi: 10.1001/jamadermatol.2013.927. PMID 23560296